CLINICAL TRIAL: NCT00983840
Title: Family Eats:Cancer Prevention for Families
Acronym: Family Eats
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Karen Cullen, Associate professor, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 124505-01A1; CA124505-01A1
Record Dates: First submitted 2009-07-30; First posted 2009-09-24 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: diet; African-American families; web-based

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Eats (Experimental): 8-session program on health eating
  Interventions: Other: Family Eats
- Family eats- plain (Active Comparator): Family eats without role model stories and goal setting
  Interventions: Other: Family Eats

INTERVENTIONS:
Other: Family Eats — 8-session web-based program on healthy eating for African American families

SUMMARY:
Poor diets lead to weight problems, and may increase cancer risk. Cancers may develop over a long period of time, with some possibly initiating in childhood. Therefore, promoting healthy diets and preventing excess weight gain during childhood could be cancer protective. Families influence children's dietary behaviors by their actions and controlling the home food environment. The internet provides family access to interventions with the convenience of the home. An eight-session interactive web-based program promoting a healthy home food environment for African-American families with 9-12 year old daughters (Family Eats) was previously developed and tested. This study tests whether the Family Eats web program improves diet and weight outcomes among 320 African-American families with 8-12 year old children. This important study will pioneer a new channel for behavior change intervention with African-American families and holds the promise of reaching large numbers of children and their families, enabling all to adopt healthy eating behaviors and achieve energy balance and reduce cancer risks.

DETAILED DESCRIPTION:
Although the burden of cancer is high among individuals of all ethnicities, ethnic differences in cancer incidence and mortality exist. African-Americans experience a higher incidence of certain cancers compared with the White population, with mortality rates at least 40% higher than other populations. Obesity, high fat, and low fruit (F) and vegetable (V) intakes increase cancer risks. Cancers may develop over a long period of time, with some possibly initiating in childhood; therefore, promoting FV and preventing excess weight gain during childhood could be cancer protective. Families influence children's dietary behaviors by direct modeling of dietary behaviors, parenting skills around food, and controlling the home food environment. However, few intervention studies have focused on family influences on dietary behaviors, particularly among ethnic minority groups which may differ in cultural and other aspects of family functioning. Unfortunately, low participation rates for community-based family interventions suggest that alternate intervention delivery systems be investigated. The internet provides family access within the convenience of the home. In a previous R21 application, the Principal Investigator developed an eight-session interactive web-based program promoting a healthy home food environment for African-American families with 9-12 year old daughters (Family Eats). Family Eats was evaluated for feasibility and changes in mediating variables were obtained. This proposal will test the efficacy of the Family Eats web program to improve FV and dietary fat behavior and weight outcomes among 320 AA families with 8-12 year old children. This important study will pioneer a new channel for behavior change intervention with African-American families and holds the promise of reaching large numbers of children and their families, enabling all to adopt healthy eating behaviors and achieve energy balance and reduce cancer risks.

ELIGIBILITY:
Inclusion Criteria:

* African -American families with 8-10 year old children
* Home computer with dsl line

Exclusion Criteria:

* Parents or children who report a medically prescribed diet, identified through a pre-screening questionnaire, will be excluded because these mothers may have received prior dietary counseling and have increased motivation for making dietary changes.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2009-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Diet (fruit, vegetables, sweetened beverages, fat and calories) | baseline, post and 6 months

SECONDARY OUTCOMES:
BMI | baseline, post and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen W Cullen, DrPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Children's Nutrition Research Center, Houston, Texas, United States